CLINICAL TRIAL: NCT01641250
Title: Open Label, Multicenter, Dose Escalation Phase 1a/b Study of RO5429083, Administered as Intravenous Infusion Alone or in Combination With Cytarabine in Patients With Acute Myelogenous Leukemia (AML).
Brief Title: A Study of RO5429083 Alone or in Combination With Cytarabine in Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28085; 2012-001027-12 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Myelogenous Leukemia, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

ARMS (2):
- Part A: RO5429083 (Experimental)
  Interventions: Drug: RO5429083
- Part B: RO5429083 + cytarabine (Experimental)
  Interventions: Drug: RO5429083; Drug: cytarabine

INTERVENTIONS:
Drug: RO5429083 — Multiple escalating doses
Drug: cytarabine — 1000 mg/m2 iv daily for 5 consecutive days, up to 4 cycles
  Arms: Part B: RO5429083 + cytarabine

SUMMARY:
This multi-center, open-label study will evaluate the safety, pharmacokinetics, pharmacodynamics and efficacy of RO5429083 alone and in combination with cytarabine in patients with acute myelogenous leukemia. In Part A, patients will receive multiple escalating doses of RO5429083 intravenously. In Part B, patients will receive RO5429083 plus up to 4 cycles of cytarabine (1000 mg/m2 iv daily for 5 consecutive days). Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed, acute myelogenous leukemia (all subtypes except acute promyelotic leukemia) according to WHO criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* All non-hematological adverse events of any prior chemotherapy, surgery, or radiotherapy must have resolved to NCI-CTC AE Grade < 2, except alopecia
* Adequate hepatic and renal function
* Patient must be willing to submit blood and bone marrow samples for PK and PD analyses and exploratory biomarkers

Exclusion Criteria:

* Patients receiving any other investigational or commercial agents or therapies administered with the intention to treat their malignancy within 14 days of first receipt of study drug, with the exception of hydroxyurea
* History of allergic reactions attributed to components of cytarabine and/or the formulated product
* Current evidence of CNS leukemia
* Increased QTc interval (QTc > 470 ms), baseline resting bradycardia < 45 beats per minute, or baseline resting tachycardia < 100 beats per minute
* Family history of long QT syndrome or other risk factors for torsades de pointes, and/or the use of concomitant medications that prolong QT/QTc interval
* Uncontrollable intercurrent illness
* Pregnant or breast-feeding women
* HIV-positive patients receiving anti-retroviral therapy

  * Patients who refuse to potentially receive blood products and/or have a hypersensitivity to blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events (including maximum tolerated dose/optimal biological dose) | approximately 24 months

SECONDARY OUTCOMES:
Clinical response according to hematologic malignancy assessments | approximately 24 months
Pharmacokinetics o RO5429083 alone and in combination with cytarabine: Area under the concentration-time curve (AUC) | Pre-dose and up to 96 hrs post-dose
Pharmacokinetics of cytarabine in combination with RO5429083: Area under the concentration-time curve (AUC) | Pre-dose and up to 24 hrs post-dose, Cycles 1 and 3
Pharmacodynamics: Biomarker levels in blood/bone marrow | Pre-dose and up to 96 hrs post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- France (4):
  - Marseille
  - Nantes
  - Paris
  - Toulouse
- Germany (3):
  - Aachen
  - Hamburg
  - Ulm
- Bologna, Emilia-Romagna, Italy